CLINICAL TRIAL: NCT02090608
Title: Paricalcitol in Fabry Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Eleonora Riccio, MD, Federico II University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCT-FD
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-01

CONDITIONS: Fabry Disease; Proteinuria
MeSH Terms: conditions — Fabry Disease; Proteinuria | interventions — paricalcitol

ARMS (1):
- Paricalcitol (Experimental): In patients identified by the inclusion criteria, data will be collected at baseline , during administration of oral Paricalcitol (PCT) (after 1, 3 and 6 months), and three months after PCT withdrawal. PCT will administered at dosage of 1 mcg/day; this dosage was chosen as it is not associated with excessive decline of parathyroid hormone (PTH) levels in most patients
  Interventions: Drug: Paricalcitol

INTERVENTIONS:
Drug: Paricalcitol — Paricalcitol was administered at the dose of 1 mcg/die

SUMMARY:
Proteinuria is the predominant risk factor for renal disease progression in Fabry disease (FD). When urine protein excretion is controlled to <0.50 g/24 hr, the rate loss of glomerular filtration rate (GFR) is not significantly different from 0. However, enzyme replacement therapy (ERT) alone does not decrease proteinuria and it has been recommended that patients receiving ERT also receive anti Renin-Angiotensin-System (RAS) therapy. Emerging evidences show that paricalcitol (PCT) reduces proteinuria in presence of intensified inhibition of RAS; however, there is no evidence in FD. The aim of this study is to evaluate the antiproteinuric effect of PCT in FD patients with proteinuria >0.50 g/24 hr persisting despite the ERT and anti-RAS therapy titrated to maximum tolerated dosage.

ELIGIBILITY:
Inclusion Criteria:

* genetically proven FD
* stable dose of ERT for at least 12 months
* stable dose of ACEi or ARB titrated to maximum tolerated dosage for at least 6 months
* persistent proteinuria >0.50 g/24 h despite the use of ERT and ACEi/ARBs in 2 consecutive samples within 12 weeks

Exclusion Criteria:

* steroid/immunosuppressive treatment or glomerular filtration rate change >30% in the past 3 months
* PTH levels <20 pg/mL
* serum phosphorus >5.0 mg/dL
* serum calcium (adjusted for albumin) >10.0 mg/dL
* active malignancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Effect of paricalcitol on proteinuria reduction | 6 months
  Fourteen Fabry patients will be selected and studied in the first six months of add-on oral PCT (1 mcg/day) and, in order to verify the dependence of proteinuria reduction on PCT, three months after drug withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: eleonora riccio, md, Principal Investigator — Federico II University
Locations (1):
- federico II university, department of nephrology, Naples, Naples, Italy